CLINICAL TRIAL: NCT02489903
Title: A Phase II Study of RRx-001 in Platinum Refractory/Resistant Small Cell Carcinoma, EGFR TKI Resistant EGFR+ T790M Negative Non-Small Cell Lung Cancer, High Grade Neuroendocrine Tumors and Resistant/Refractory Ovarian Cancer Prior to Re-administration of Platinum Based Doublet Regimens (QUADRUPLE THREAT)
Brief Title: RRx-001 in Lung Cancer, Ovarian Cancer and Neuroendocrine Tumors Prior to Re-administration of Platinum Based Doublet Regimens (QUADRUPLE THREAT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EpicentRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRx001-211-01
Record Dates: First submitted 2015-06-29; First posted 2015-07-03 (Estimated); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Small Cell Carcinoma; Carcinoma, Non-Small-Cell Lung; Neuroendocrine Tumors; Ovarian Epithelial Cancer
Keywords: Epigenetics; resensitization; Platinum doublets; lung cancer; Ovarian epithelial cancer
MeSH Terms: conditions — Carcinoma, Small Cell; Carcinoma, Non-Small-Cell Lung; Neuroendocrine Tumors; Carcinoma, Ovarian Epithelial; Lung Neoplasms | interventions — RRx-001; Cisplatin; Etoposide; Carboplatin; Irinotecan; Vinorelbine; liposomal doxorubicin; Gemcitabine; taxane; Paclitaxel; 130-nm albumin-bound paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Small Cell Lung Cancer (Arm 1) (Experimental): RRx-001 weekly for 3 weeks followed by up to 4 cycles of carboplatin or cisplatin plus etoposide and then RRx-001 and carboplatin or cisplatin (for patients with stable disease (SD) or better at discontinuation of platinum).
  Interventions: Drug: RRx-001; Drug: Cisplatin; Drug: Etoposide; Drug: Carboplatin
- Small Cell Lung Cancer (Arm 2) (Active Comparator): Carboplatin or cisplatin plus etoposide or irinotecan or vinorelbine until progression or intolerable toxicity
  Interventions: Drug: Cisplatin; Drug: Etoposide; Drug: Carboplatin; Drug: Irinotecan; Drug: Vinorelbine
- Non Small Cell Lung Cancer (Experimental): RRx-001 weekly for 3 weeks followed by up to 6 cycles of cisplatin or carboplatin plus paclitaxel or nab-paclitaxel or pemetrexed and then RRx-001 maintenance (for patients with stable disease or better at discontinuation of platinum).
  Interventions: Drug: RRx-001; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-Paclitaxel; Drug: Pemetrexed
- Neuroendocrine tumors (Experimental): RRx-001 weekly until progression followed by up to 6 cycles of carboplatin or cisplatin plus etoposide and then RRx-001 maintenance (for patients with stable disease or better at discontinuation of platinum).
  Interventions: Drug: RRx-001; Drug: Cisplatin; Drug: Etoposide; Drug: Carboplatin
- Ovarian epithelial cancer (Arm 1) (Experimental): RRx-001 weekly for 2 weeks followed by 2 cycles of Carboplatin chemotherapy and then RRx-001/Carboplatin maintenance (for patients with stable disease or better at discontinuation of platinum).
  Interventions: Drug: RRx-001; Drug: Carboplatin
- Ovarian epithelial cancer (Arm 2) (Active Comparator): Carboplatin, Etoposide, Doxil, Gemcitabine or Vinorelbine or Taxane until progression or intolerable toxicity
  Interventions: Drug: Etoposide; Drug: Carboplatin; Drug: Vinorelbine; Drug: Doxil; Drug: Gemcitabine; Drug: Taxane

INTERVENTIONS:
Drug: RRx-001
  Arms: Neuroendocrine tumors; Non Small Cell Lung Cancer; Ovarian epithelial cancer (Arm 1); Small Cell Lung Cancer (Arm 1)
Drug: Cisplatin
  Arms: Neuroendocrine tumors; Non Small Cell Lung Cancer; Small Cell Lung Cancer (Arm 1); Small Cell Lung Cancer (Arm 2)
Drug: Etoposide
  Arms: Neuroendocrine tumors; Ovarian epithelial cancer (Arm 2); Small Cell Lung Cancer (Arm 1); Small Cell Lung Cancer (Arm 2)
Drug: Carboplatin
Drug: Irinotecan
  Arms: Small Cell Lung Cancer (Arm 2)
Drug: Vinorelbine
  Arms: Ovarian epithelial cancer (Arm 2); Small Cell Lung Cancer (Arm 2)
Drug: Doxil
  Arms: Ovarian epithelial cancer (Arm 2)
Drug: Gemcitabine
  Arms: Ovarian epithelial cancer (Arm 2)
Drug: Taxane
  Arms: Ovarian epithelial cancer (Arm 2)
Drug: Paclitaxel
  Arms: Non Small Cell Lung Cancer
Drug: Nab-Paclitaxel
  Arms: Non Small Cell Lung Cancer
Drug: Pemetrexed
  Arms: Non Small Cell Lung Cancer

SUMMARY:
This study is designed to explore the potential of the epigenetic agent RRx-001 to sensitize patients who previously received and now have failed a platinum based doublet regimen. RRx-001 is administered with autologous blood once weekly followed by or in combination with reintroduction of platinum-based doublet therapy.

DETAILED DESCRIPTION:
This is an open label, four 'cohort' study for administration of RRx-001 with autologous blood once weekly followed by or in combination with reintroduction of platinum-based doublet therapy according to the treatment schedule listed below. Small cell carcinoma and ovarian cohort participants will be randomized to 1 of 2 treatment arms, respectively. Neuroendocrine and NSCLC patients will be enrolled to single arms.

Participants with SCC will receive one of the following; RRx-001 followed by platinum doublet chemotherapy or platinum based chemotherapy alone. HGNEC, RRx-001 followed by platinum doublet chemotherapy. NSCLC, RRx-001 followed by platinum doublet chemotherapy. Participants with Platinum Refractory/Resistant Ovarian and MMMT will receive one of the following, RRx-001 followed by platinum doublet chemotherapy or chemotherapy alone.

Approximately 213 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria

* Patients must have histologically or cytologically confirmed advanced or metastatic:

  * Resistant/Refractory Small Cell Carcinoma (SCC) patients in 3rd line or beyond that have previously received platinum or patients in 2nd line with platinum-refractory or platinum-resistant disease
  * EGFR mutated non-small cell lung cancer (NSCLC) that has previously received a first line platinum doublet and all applicable EGFR TKIs
  * Epithelial Ovarian Cancer (EOC), fallopian tube or primary peritoneal cancer and Malignant Mixed Mullerian Tumor (MMMT) of the ovary or uterus. Excludes other non-epithelial ovarian tumors and ovarian tumors with low malignant potential. Patients must have previously received a platinum based regimen for advanced/metastatic disease or have platinum resistant or refractory disease defined as relapse within 6 months. EOC - specific criteria: Patients who progress or have stable disease during first-line treatment or who relapse within 1 month are considered to be 'platinum-refractory'. Patients who respond to primary treatment and relapse within 6 months are considered 'platinum-resistant', and patients who relapse more than 6 months after completion of initial therapy are characterized as 'platinum-sensitive'. Patients who relapse 6-12 months following the end of their initial regimen are classified as 'partially sensitive'. Platinum sensitive patients may be enrolled but must have failed or declined all other lines of FDA approved therapy
  * High-Grade Neuroendocrine Carcinoma (HGNEC), any organ of origin, including a pathology of neuroendocrine features, in patients previously been treated with chemotherapy Although neuroendocrine tumors may be classified differently based on organ of origin, in the context of this protocol they are defined as high grade on the basis of either

    1. Aggressive clinical behavior requiring previous treatment with chemotherapy even if histologic features such as the Ki67 index or mitotic rate corresponds with low or intermediate grade.
    2. Histologic features: (a) Neuroendocrine tumors of lung origin are considered high grade if in any part of the tumors, there are >10 mitoses/2mm2 or 10 high power field (HPF). Large zones of necrosis are usually present. This includes small cell lung carcinoma and large cell neuroendocrine lung carcinoma. [SCLC will not enroll in the HGNEC cohort.] (b)Neuroendocrine tumors of gastroenteropancreatic origin are considered high grade if in any part of the tumors there are either >20 mitoses/2mm2 or 10 high power field (HPF) OR Ki67.
* Radiographically measurable disease by RECIST v1.1
* A washout period of 3-weeks from last treatment.
* Patients must have previously received a platinum based regimen for advanced/metastatic disease and progressed or have platinum resistant or refractory disease defined as relapse within 6 months.
* Age ≥18 years.
* Life expectancy of ≥12 weeks.
* ECOG performance status 0-2.
* Participants must have adequate organ and marrow function as defined below both prior to administration of RRx-001 and prior to administration of platinum doublet based regimen:

  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL (non-transfused platelet count)
  * Hemoglobin ≥9 g/dL (transfused Hgb allowed)
  * Creatinine ≤1.5 x the upper limit of normal
  * Total bilirubin ≤2.0 x the upper limit of normal or <3.0 xULN if patient has a history of Gilbert's syndrome
  * AST (SGOT)/ALT (SGPT) ≤5 X institutional upper limit of normal if with liver metastases; ≤2.5 X ULN if no liver metastases
* Patient must consent to the access, review and analysis of previous medical and cancer history, including tumor archival tissue (if available) and imaging data by the sponsor or a third party nominated by the sponsor.
* Ability to understand and sign a written informed consent document.
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.

  * Note: A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: Has not undergone a hysterectomy or bilateral oophorectomy; or Has not been postmenopausal for at least 12 consecutive months

Exclusion Criteria

* Receiving concurrent investigational therapy
* Symptomatic central nervous system metastasis (e.g., patients requiring increasing doses of steroids)
* History of needing to permanently discontinue prior platinum doublet-based regimen for toxicity (e.g., cisplatin causing renal impairment, ototoxicity, or severe neuropathy).
* Known severe hypersensitivity to the platinum agent (i.e., carboplatin or cisplatin) or prior partner of platinum agent (i.e., etoposide for SCC and HGNEC; nab-paclitaxel, paclitaxel, or pemetrexed for NSCLC; paclitaxel, pegylated liposomal doxorubicin, docetaxel or gemcitabine for ovarian) planned for the platinum therapy period. If the patient has had prior hypersensitivity reaction to the drug partner of platinum, a patient may enroll as long as it is acceptable to treat with platinum and one of the alternative chemotherapy partner agents.
* Any significant medical diseases or conditions, as assessed by the investigators and sponsor that would substantially increase the medical risks of participating in this study (i.e., uncontrolled diabetes, NYHA II-IV congestive heart failure, myocardial infarction within 6 months of study, severe chronic pulmonary disease or active uncontrolled infection, uncontrolled or clinically relevant pulmonary edema).
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Oronsky, MD, PhD, Study Director — EpicentRx, Inc.
Locations (10):
- United States (10):
  - Stanford University, Palo Alto, California
  - VA Connecticut Cancer Center, West Haven, Connecticut
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Baptist Health, Lexington, Kentucky
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Henry Ford Allegiance Health, Jackson, Michigan
  - Washington University, St Louis, Missouri
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Virginia Cancer Specialists, Fairfax, Virginia
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Derived] Tomita Y, Oronsky B, Abrouk N, Cabrales P, Reid TR, Lee MJ, Yuno A, Baker J, Lee S, Trepel JB. In small cell lung cancer patients treated with RRx-001, a downregulator of CD47, decreased expression of PD-L1 on circulating tumor cells significantly correlates with clinical benefit. Transl Lung Cancer Res. 2021 Jan;10(1):274-278. doi: 10.21037/tlcr-20-359. PMID 33569311
- [Derived] Morgensztern D, Rose M, Waqar SN, Morris J, Ma PC, Reid T, Brzezniak CE, Zeman KG, Padmanabhan A, Hirth J, I Spira A, Trepel JB, Padda SK. RRx-001 followed by platinum plus etoposide in patients with previously treated small-cell lung cancer. Br J Cancer. 2019 Jul;121(3):211-217. doi: 10.1038/s41416-019-0504-8. Epub 2019 Jun 24. PMID 31231122

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 13 academic medical centers between June 2015 and October 2020. The first participant first visit was June 12, 2015 and the last patient last visit was October 8, 2020.
Pre-assignment Details: 139 participants provided consent. 118 patients consented under Amendment 01-09. 21 patients were consented on Amendment 10 with 13 randomized in the study.
  A total of 92 patients under Amendment 01-09 and 13 patients under Amendment 10, combined 107 patients.
Groups:
- RRx-001 + Platinum Doublet (A01-09): 4mg RRx-001 once weekly (QW) until progression, followed by up to 6 cycles of platinum doublet chemotherapy
- RRx-001 + Platinum + RRx-001 (A10): RRx-001 weekly for 3 weeks followed by up to 6 cycles of platinum doublet chemotherapy and then RRx-001 maintenance (for patients with stable disease (SD) or better at discontinuation of platinum).
- Investigator's Choice (A10): Standard of Care Investigator's Choice Control Arm, treatment options of one of the following: carboplatin, etoposide, doxil, gemcitabine, vinorelbine or taxane treatments until progression or intolerable toxicity
- Screening (Pre-Randomization) (A10): Subjects were screened and did not get Randomized
Period: Screening
Arm/Group | RRx-001 + Platinum Doublet (A01-09) | RRx-001 + Platinum + RRx-001 (A10) | Investigator's Choice (A10) | Screening (Pre-Randomization) (A10)
Started | 118 | 0 | 0 | 21
Completed | 94 | 0 | 0 | 13
Not Completed | 24 | 0 | 0 | 8
Not completed — Screen Failure | 24 | 0 | 0 | 8
Period: Randomized and Received Treatment
Arm/Group | RRx-001 + Platinum Doublet (A01-09) | RRx-001 + Platinum + RRx-001 (A10) | Investigator's Choice (A10) | Screening (Pre-Randomization) (A10)
Started | 94 | 11 | 2 | 0
Completed | 75 | 7 | 2 | 0
Not Completed | 19 | 4 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Baseline Drop Out | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 0 | 0
Not completed — Death | 10 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population comprises all subjects who are randomized and received at least 1 dose of study drug and will be used for all analyses of safety. Analysis is based on actual treatment group
Groups:
- Total: Total of all reporting groups
Arm/Group | RRx-001 + Platinum Doublet (A01-09) | RRx-001 + Platinum + RRx-001 (A10) | Investigator's Choice (A10) | Total
Number analyzed (Participants) | 94 | 11 | 2 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (11.3) | 61.3 (6.1) | 75.0 (2.8) | 61.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 8 | 0 | 56
  Male | 46 | 3 | 2 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 88 | 10 | 2 | 100
  Unknown or Not Reported | 3 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 1 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 0 | 3
  Black or African American | 10 | 0 | 0 | 10
  White | 74 | 9 | 2 | 85
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 94 | 11 | 2 | 107

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: From the time from enrollment until the time of death from any cause or last follow-up. Patients will be followed clinically as outlined in the treatment schedule and will be followed off study for death.
Time Frame: From start of treatment through death for up to 64 months from Start of Treatment.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | RRx-001 + Platinum Doublet (A01-09) | RRx-001 + Platinum + RRx-001 (A10) | Investigator's Choice (A10)
Number analyzed (Participants) | 89 | 10 | 2
Months | 6.85 [5.80 to 8.62] | 7.6 [5.00 to NA] — insufficient number of participants with events | 7.5 [3.00 to NA] — insufficient number of participants with events

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) will be defined as the proportion of patients with a CR or a PR per RECIST v1.1 based upon the best response as assessed; confirmation of response was not required, assessed up to 49 months.
Time Frame: Assessed up to 49 months
Measure: Count of Participants; unit: Participants
Arm/Group | RRx-001 + Platinum Doublet (A01-09) | RRx-001 + Platinum + RRx-001 (A10) | Investigator's Choice (A10)
Number analyzed (Participants) | 89 | 10 | 2
Participants | 32 | 3 | 1

3. Secondary Outcome: Disease Control Rate (DCR)
Description: The percentage of patients who have achieved complete response, partial response and stable disease (as per RECIST v1.1), assessed up to 49 months.
Time Frame: Assessed up to 49 months
Measure: Count of Participants; unit: Participants
Arm/Group | RRx-001 + Platinum Doublet (A01-09) | RRx-001 + Platinum + RRx-001 (A10) | Investigator's Choice (A10)
Number analyzed (Participants) | 89 | 10 | 2
Participants | 42 | 8 | 2

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) will be defined as the elapsed time from the from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 49 months.
Time Frame: Assessed up to 49 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RRx-001 + Platinum Doublet (A01-09) | RRx-001 + Platinum + RRx-001 (A10) | Investigator's Choice (A10)
Number analyzed (Participants) | 89 | 10 | 2
months | 5.87 [4.46 to 7.54] | 6.50 [NA to NA] — insufficient number of participants with events | 12 [NA to NA] — insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Adverse Events were collected beginning at baseline through end of treatment (28 days after last dose of study drug), up to 64 months. All-Cause Mortality was assessed from baseline through 28 days after last dose of study drug.
Description: All Serious Adverse Events are reported irregardless of attribution. Adverse events are reported for related to study treamtent. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 is used to grade adverse events.
Arm/Group | RRx-001 + Platinum Doublet (A01-09) | RRx-001 + Platinum + RRx-001 (A10) | Investigator's Choice (A10)
All-Cause Mortality (participants affected / at risk) | 89/89 | 10/10 | 2/2
Serious Adverse Events (participants affected / at risk) | 55/89 | 6/10 | 2/2
Other Adverse Events (participants affected / at risk) | 89/89 | 10/10 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RRx-001 + Platinum Doublet (A01-09) (N=89) | RRx-001 + Platinum + RRx-001 (A10) (N=10) | Investigator's Choice (A10) (N=2)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Supraventricular Tachycardia (SVT) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cushing's Syndrome (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Abdominal Pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Duodenal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obstruction Gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Death (General disorders) | 6 (6) | 0 (0) | 0 (0)
Generalized Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Coronavirus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Spinal Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Bladder Outlet Obstruction (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Drug Reaction with Eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Inferior Vena Cava Syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic Venous Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superior Vena Cava Syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RRx-001 + Platinum Doublet (A01-09) (N=89) | RRx-001 + Platinum + RRx-001 (A10) (N=10) | Investigator's Choice (A10) (N=2)
Anaemia (Blood and lymphatic system disorders) | 12 (27) | 8 (8) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 9 (13) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 11 (18) | 0 (0) | 0 (0)
Tumour pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (12) | 4 (6) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 9 (12) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 20 (23) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (25) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (13) | 2 (2) | 0 (0)
Fatigue (General disorders) | 18 (35) | 4 (7) | 1 (1)
Infusion related reaction (Investigations) | 18 (18) | 4 (7) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 (12) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (13) | 1 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 9 (11) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 8 (11) | 2 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT02489903/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT02489903/ICF_001.pdf